CLINICAL TRIAL: NCT04538859
Title: A Prospective Study of Factors Related to Exacerbation and Mortality of Non-cystic Fibrosis Bronchiectasis in Hong Kong
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Susanna SS Ng, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: ProBronchiectasis/2019
Record Dates: First submitted 2020-08-31; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bronchiectasis is associated with repeated exacerbations which occurs at rates of 1.5-6.5 per patients per year, and are associated with an increased risk of admission and readmission to hospital, and high health care costs. In a local study carried out more than 10 years ago, idiopathic disease dominates and patients with bronchiectasis are mainly female with high hospitalization and mortality rates; 21.9 cases per 100,000 and 2.7 cases per 100,000 respectively. Moreover, exacerbation characterized by increases in symptoms requiring antibiotic treatment is associated with disease progression and significant mortality. Updated prevalence of this disease with the characteristics of etiology, clinical presentation and outcomes are needed to guide further management plan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older
2. Clinically stable for at least 4 weeks prior to enrollment (defined as no symptoms of exacerbation, no requirement for supplemental antibiotic therapy)
3. Diagnosis of bronchiectasis defined by high-resolution computed tomography scan

Exclusion Criteria:

1. History of cystic fibrosis; hypogammaglobulinemia; allergic bronchopulmonary aspergilosis
2. Those who are unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study of patients. We propose to recruit consecutive patients who are under care of the Respiratory Clinic at the Prince of Wales Hospital with the diagnosis of bronchiectasis defined by high-resolution Computed Tomography scan. Patients who recover from a recent admission the Prince of Wales Hospital with exacerbation of bronchiectasis will also be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-30 (Actual); Primary Completion 2027-08-29 (Estimated); Study Completion 2027-08-29 (Estimated)

PRIMARY OUTCOMES:
Number of bronchiectasis exacerbation | 5 years

SECONDARY OUTCOMES:
Mortality rate | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong, Hong Kong, Please Select, Hong Kong

IPD SHARING:
Plan to Share IPD: No